CLINICAL TRIAL: NCT04233346
Title: A Phase II Multi-center, Randomized, Open-label Study of Ponatinib in Chinese Patients With Chronic Myeloid Leukemia Who Have Failed Prior TKIs or With T315I Mutation, or Ph+ALL Who Have Failed Prior TKIs or With T315I Mutation
Brief Title: The Study for CML Who Failed Prior TKIs or With T315I Mutation or Ph+ ALL Who Failed Prior TKIs or With T315I Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 297-403-00003
Record Dates: First submitted 2019-12-31; First posted 2020-01-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; ponatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ponatinib 30mg (Experimental): 50% CML patients will be treated with 30mg/day ponatinib，the treatment will up to 60 months
  Interventions: Drug: Ponatinib 30mg OD
- Ponatinib 45mg (Experimental): 50% CP-CML patients will be randomized 45 mg dose group . Other patients (with AP-CML, BP-CML, Ph+ ALL) will only be assigned to 45 mg dose group(30 patients). The treatment will up to 60 months.
  Interventions: Drug: Ponatinib 45mg OD

INTERVENTIONS:
Drug: Ponatinib 30mg OD — Ponatinib 30mg OD
  Arms: Ponatinib 30mg
Drug: Ponatinib 45mg OD — Ponatinib 45mg OD
  Arms: Ponatinib 45mg

SUMMARY:
This protocol will allow ponatinib with refractory Chronic Myeloid Leukemia or Ph+ Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and efficacy of ponatinib in patients with chronic myeloid leukemia (CML) in chronic phase (CP), accelerated phase (AP) or blast phase (BP) or with Ph positive (Ph+) acute lymphoblastic leukemia (ALL) who either are resistant or intolerant to either dasatinib or nilotinib, or have the T315I mutation.

ELIGIBILITY:
Inclusion Criteria:

For CP-CML patients：

1. Patients with CP-CML

   Patients must either meet criterion 2 or 3:
2. Be previously treated with and resistant or intolerant to either Dasatinib or Nilotinib:
3. Develop the T315I mutation after any TKI therapy;
4. Must be ≥18 years old.
5. Provide written informed consent.
6. Eastern Cooperative Oncology Group performance status ≤ 2.
7. Minimum life expectancy of 3 months or more.
8. Adequate renal function
9. Adequate hepatic function
10. Normal pancreatic status
11. Normal QTc interval on screening electrocardiogram (ECG) evaluation under resting state, defined as QTc of ≤ 450 ms in males or ≤ 470 ms in females.

For AP/BP-CML and ALL patients：

1. Patients with AP-CML and BP-CML or Ph+ ALL
2. Other inclusions are the same with No.2-No.11 of CP-CML patients

Exclusion Criteria:

For CP-CML patients：

1. Received TKI therapy within 7 days prior to receiving the first dose of Ponatinib, or have not recovered (> grade 2 by NCI CTCAE v5.0) from AEs (except alopecia) due to agents previously administered.
2. Received other therapies (excluding hydroxyurea) as follows:

   Received interferon, cytarabine, or immunotherapy within 14 days, or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy within 28 days prior to receiving the first dose of Ponatinib.
3. Underwent autologous or allogeneic stem cell transplant < 60 days prior to receiving the first dose of Ponatinib;
4. Take medications that are known to be associated with Torsades de Pointes or QT interval prolongation.
5. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
6. Have previously been treated with Ponatinib or its analogues (including drug substance).
7. Patients with CP-CML are excluded if they are in CCyR.
8. Have active central nervous system (CNS) disease, as evidenced by cytology or pathology.
9. Have significant, uncontrolled, or active heart/brain/peripheral vascular diseases
10. Have a significant bleeding disorder unrelated to CML
11. Have a history of pancreatitis or alcohol abuse
12. Severely increased hypertriglyceridemia (triglycerides ≥ 5.6 mmol/L).
13. Have malabsorption syndrome or other gastrointestinal illness that could affect absorption of orally administered Ponatinib.
14. Have been diagnosed with another primary malignancy within the past 3 years (except for non-melanoma skin cancer, cervical cancer in situ, or controlled prostate cancer, which are allowed within 3 years).
15. Are pregnant or lactating.
16. Underwent major surgery (with the exception of minor surgical procedures, such as catheter placement or BM biopsy) within 14 days prior to first dose of Ponatinib.
17. Infectious diseases test showed anti-HIV (+) or anti-HCV (+) or HbsAg (+) or TP (+).
18. Suffer from any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the safety of the study drug.
19. Have hypertension (diastolic blood pressure ≥ 90 mmHg and/or systolic blood pressure ≥ 140 mm Hg).
20. Taken herbal preparations or related over-the-counter preparations containing Chinese herbal ingredients within 2 weeks prior to the first dose of Ponatinib.
21. Any subject who is not suitable for the study in the opinion of the investigator.

For AP/BP-CML and ALL patients：

1. Received TKI therapy within 7 days prior to receiving the first dose of Ponatinib, or have not recovered (> grade 2 by NCI CTCAE v.5.0) from AEs (except alopecia) due to agents previously administered.
2. Received other therapies (excluding hydroxyurea) as follows:

   For AP-CML patients, received interferon, cytarabine, or immunotherapy within 14 days, or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy within 28 days prior to receiving the first dose of Ponatinib.

   For BP-CML patients, received chemotherapy within 7 days prior to the first dose of Ponatinib. Otherwise, 2a applies.

   For Ph+ ALL patients, received corticosteroids within 24 hours before the first dose of Ponatinib; otherwise, 2a applies.
3. Underwent autologous or allogeneic stem cell transplant < 60 days prior to receiving the first dose of Ponatinib.
4. Take medications that are known to be associated with Torsades de Pointes or QT interval prolongation.
5. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
6. Have previously been treated with Ponatinib or its analogues (including drug substance).
7. Patients with AP-CML, BP-CML, or Ph+ ALL are excluded if they are in MaHR.
8. Patients with AP-CML, BP-CML, or Ph+ ALL are excluded if a baseline BM aspirate adequate for cell count and differential report is not available.
9. Have active central nervous system (CNS) disease as evidenced by cytology or pathology for AP-CML, BP-CML, or Ph+ ALL.
10. Have significant, uncontrolled, or active cardiovascular disease.
11. Have a significant bleeding disorder unrelated to CML or Ph+ ALL.
12. Other exclusions are the same with No.11-No.21 of CP-CML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MCyR(Major Cytogenetic Response) of CP-CML patients | 12 months
  To confirm the efficacy of Ponatinib in Chinese patients with CML who have failed Dasatinib or Nilotinib or with T315I mutation, or Ph+ ALL who have failed prior TKIs or with T315I mutation as evidenced by cytogenetic responses
MaHR(Major Hematologic Response) of AP-CML, BP-CML and Ph+ ALL patients by 6 months | 6 months
  To confirm the efficacy of Ponatinib in Chinese patients with CML who have failed Dasatinib or Nilotinib or with T315I mutation, or Ph+ ALL who have failed prior TKIs or with T315I mutation as evidenced by hematology responses

SECONDARY OUTCOMES:
Duration of response | Up to 5 years
  Assessment in the total patient population
Progression-free survival (PFS) | Up to 5 years
  Assessment in the total patient population
Overall survival (OS) | Up to 5 years
  Assessment in the total patient population
Time to response (TTR) | Up to 5 years
  Assessment in the total patient population
Adverse events | Up to 5 years
  Number of participants with adverse events as assessed by CTCAE v5.0
EORTC QLQ-C30 (version 3) | Up to 5 years
  EORTC QLQ-C30 (version 3) score ranges from 1 to 4 or 1 to 7, A higher score represents a severer impressions or a best applies of patients.
Maximum Plasma Concentration [Cmax] | Up to 3 months
  Plasma concentration-time data for the population PK study

CONTACTS AND LOCATIONS:
Overall Officials: Juma Paty, Director, Study Director — OBRI
Locations (14):
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shenzhen Second People's Hospital, Shenzhen, Shenzhen
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - 1st affiliated hospital, Peking University, Beijing
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin

IPD SHARING:
Plan to Share IPD: No